CLINICAL TRIAL: NCT05365139
Title: Diagnostic Tools for Identifying Prolonged Grief: Development and Validation of the First Clinical Diagnostic Interview for Assessing Prolonged Grief Disorder With the ICD 11 Criteria and DSM-5 Tr Criteria.
Brief Title: Diagnostic Tools for Identifying Prolonged Grief
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Maja O'Connor, Professor, University of Aarhus
Other Study IDs: 35880 Aarhus University
Record Dates: First submitted 2021-12-06; First posted 2022-05-09 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Prolonged Grief Disorder
Keywords: PGD; prolonged grief disorder; clinical interview; ICD-11 PGD; DSM-5 Tr PGD
MeSH Terms: conditions — Prolonged Grief Disorder | interventions — Prostaglandins D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Structured clinical diagnostic interview for PGD (PGD-I) — Participants were administered the Structured clinical diagnostic interview for PGD (PGD-I) and screened with clinical interviews for PTSD, anxiety and depression. Whether the Aarhus PGD-scale should be answered before or after the interview was randomized.
  The PGD-I and self-report scale were readministered to 50 participants 7-14 days after the initial administration.

SUMMARY:
Development and validation of first clinical diagnostic interview for assessing Prolonged Grief Disorder (PGD) with the ICD 11 and DSM 5 Tr criteria.

DETAILED DESCRIPTION:
Development and validation of first clinical diagnostic interview for assessing Prolonged Grief Disorder (PGD) with the ICD 11 and DSM 5 Tr criteria.

Background: With WHO's introduction of PGD in the ICD 11, which will be implemented in Health Services worldwide from January 2022, there is a need to accurately diagnose people with ICD-11PGD (PGD caseness) with a valid structured clinical interview.

With ICD-11 a slightly different set of symptoms for PGD is defined as the gold standard for PGD. This standard will be used for diagnosing and understanding PGD in future research and health service. ICD-11 aims to be descriptive, e.g. provides a support for the clinicians to identify PGD by describing common reactions and symptoms of this disorder, but there is still a need to evaluate the validity of these criteria. Strict diagnostic criteria with defined numbers, combinations, and intensity of symptoms (e.g. for the use in research) are not yet defined in ICD-11 and no structured clinical interview that measure ICD-11 or the upcoming DSM 5 tr PGD has yet been developed and validated for this purpose. This means that the field currently stand without reliable ways to classify accurately who has PGD diagnosis and who has not. Without such constructs, PGD is not possible to identify, and ultimately to treat, in a validated and reliable way.

There is therefore a need to develop accurate tests that measure ICD 11 PGD, both in a structured clinical interview for use in direct meetings between patients and health service professionals and in relation to a self-report scale. The investigators already developed the Aarhus PGD scale but still need a structured clinical interview.

Aim: In this project we will

1. Develop and validate the first structured, clinical interview for ICD-11 PGD and DSM-5 Tr PGD
2. Identify a valid clinical cut-off for diagnostic PGD on The Aarhus PGD Scale.

Method:

Based on the ICD-11 and DSM 5 Tr PGD criteria and our work with the self-report scale above the investigators will develop a structured, clinical interview, The Aarhus PGD Interview, in line with the strategy used in SCID-I interviews [6]. This study will examine the content validity, the concurrent validity, the test-retest reliability and the inter-rater reliability of this interview.

After the Aarhus PGD Interview is validated, this study will compare the participant's scores on the Aarhus PGD Scale for ICD 11 and DSM 5 Tr PGD with the clinical interview as the gold standard. This will allow investigating the diagnostic test accuracy of the ICD-11 PGD scale, and to identify a valid clinical cut-off on this scale.

Perspectives: The main aim of this study is to develop and validate the first structured, clinical interview for ICD 11 and DSM 5 Tr PGD. It will provide reliable constructs to separate PGD from other, trans-diagnostic forms of complicated grief reactions such as PTSD, depression and anxiety following a loss. The ability to identify who actually has a diagnosis of PGD and are in need of treatment is crucial to be able to allocate health benefits as efficient and helpful as possible. It is also crucial in identifying the vast majority of bereaved people with normal grief reactions, and to reduce the risk of pathologizing healthy grief, which is a concern brought on by the introduction of PGD as a diagnostic entity

ELIGIBILITY:
Inclusion Criteria:

* Bereaved by the loss a loved one to death minimum 6 month ago
* 18 years or above
* The grief is still (more or less) affecting function/everyday life

Exclusion Criteria:

* Bereaved by other losses than a loved person (e.g., pet, divorce)
* 17 years or younger
* Less than 6 month ago since the loss.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Bereaved (Danish) persons who lost a loved one minimum 6 month ago.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Prolonged grief disorder (ICD-11 and DSM-TR) | 1 day
  The Aarhus PGD-interview (dichotomous scoring 0/1 (1 equals worse outcome))

SECONDARY OUTCOMES:
Post traumatic stress disorder | 1 day
  the MINI interview adapted to DSM-5 PTSD criteria (structured clinical interview, dichotomous scoring 0/1 (1 equals worse outcome))
Depression and generalized anxiety disorder | 1 day
  The Schedules for Clinical Assessment in Neuropsychiatry (SCAN) (semi-structrured clinical interview, dichotomous scoring 0/1 (1 equals worse outcome))
The Aarhus PGD-Scale | 1 day
  Self report questionnaire based on 26 5-point Likert scale items (higher scores equals worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Maja O'Connor, Principal Investigator — Aarhus Universitet
Locations (1):
- Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No